CLINICAL TRIAL: NCT01165424
Title: A Study of Long-term (12-24 Weeks) Administration of Mometasone Furoate Nasal Spray in Pediatric Subjects With Perennial Allergic Rhinitis (Protocol No. P06333)
Brief Title: A Study of Long-term Administration of Mometasone Furoate Nasal Spray in Pediatric Subjects With Perennial Allergic Rhinitis (Study P06333AM1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P06333
Record Dates: First submitted 2010-05-28; First posted 2010-07-19 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MFNS 50 μg device (Experimental): MFNS 50 μg spray device. The dose will be as follows:
  * 3 to 11 years: one spray per nostril once daily (100 μg/day) in the morning.
  * 12 to 15 years: 2 sprays per nostril once daily (200 μg/day) in the morning.
  Interventions: Drug: mometasone furoate

INTERVENTIONS:
Drug: mometasone furoate — MFNS 50 μg spray device
  * 3 to 11 years: one spray per nostril once daily (100 μg/day) in the morning.
  * 12 to 15 years: 2 sprays per nostril once daily (200 μg/day) in the morning.
  Other Names: Nasonex

SUMMARY:
Mometasone furoate nasal spray (MFNS) is a once-a-day product. This is a multi-center, open-label study of MFNS in children with perennial allergic rhinitis. MFNS will be administered to pediatric subjects (3-15 years old) with perennial allergic rhinitis at a dose of 100 to 200 μg/day (once daily) for 12 weeks. Subjects (subject's legal representatives) provided consent to continue treatment beyond 12 weeks will receive treatment for up to 24 weeks. At each clinic visit, observation of adverse events, nasal symptom scores, and nasal findings will be evaluated. The presence/absence of serious adverse events and trial procedure-related AEs will be reviewed 30 days after the end of the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having symptoms of perennial allergic rhinitis of moderate to severe degree.
* Subjects confirmed to be allergic to non-seasonal environmental antigens (e.g., house dust mite antigen).
* Male or female outpatients aged 3 to 15 years at the time of providing informed consent.

Exclusion Criteria:

* Subjects with coexisting tuberculosis or lower respiratory tract infection, or who have an acute upper respiratory tract infection or acute pharyngolaryngitis, etc. judged by the investigator to require treatment at the time of registration
* Subjects with coexisting infections or systemic mycosis for which there are no effective antibiotics
* Subjects with repeated epistaxis
* Subjects with coexisting fungal infection in nasal/sinus cavity
* Subjects with a history of hypersensitivity to steroids or ingredients of mometasone furoate nasal spray
* Subjects with severe hepatic, renal, cardiac, hematological disease, diabetes mellitus, hypertension, or other serious coexisting diseases and whose general condition is poor.
* Subjects allergic to pollen (cedar, Japanese cypress, birch, grasses, mugwort, common ragweed, etc.) for whom the pollen season coincides with the observation period

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MFNS: Mometasone furoate nasal spray (MFNS) 50 mcg device.
  Participants aged 3 to 11 years received one spray per nostril once daily (100 mcg/day) in the morning for up to 24 weeks.
  Participants aged 12 to 15 years received 2 sprays per nostril once daily (200 mcg/day) in the morning for up to 24 weeks.
Period: Overall Study
Arm/Group | MFNS
Started | 80
Completed | 76
Not Completed | 4
Not completed — Clinical adverse experiences | 1
Not completed — Laboratory adverse experiences | 1
Not completed — Did not meet entry criteria | 1
Not completed — Participant moved (relocated) | 1

BASELINE CHARACTERISTICS:
Arm/Group | MFNS
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 54
Region of Enrollment [Number; unit: Participants]
  Japan | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Adverse Drug Reactions
Time Frame: Baseline to Week 24
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | MFNS
Number analyzed (Participants) | 80
participants
  Number with Adverse Events | 76
  Number with Adverse Drug Reactions | 18

2. Secondary Outcome: Change From Baseline in the Total Nasal Symptom Score
Description: Total nasal symptom score was a composite of 4 symptoms (sneezing, rhinorrhea, nasal congestion, and nasal itching). Each symptom was scored on a scale of 0 = none, 1 = mild, 2 = moderate, and 3 = severe for a total score ranging from 0 to 12. A higher score indicates more severe symptoms.
Time Frame: Baseline and Weeks 2, 4, 8, 12, and 24 (or discontinuation)
Population: All treated participants
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MFNS
Number analyzed (Participants) | 80
units on a scale
  Change at Week 2 | -3.1 (0.3)
  Change at Week 4 | -3.9 (0.3)
  Change at Week 8 | -4.4 (0.3)
  Change at Week 12 | -4.5 (0.3)
  Change at Week 24 | -4.8 (0.3)

ADVERSE EVENTS:
Arm/Group | MFNS
Serious Adverse Events (participants affected / at risk) | 1/80
Other Adverse Events (participants affected / at risk) | 72/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MFNS (N=80)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MFNS (N=80)
Abdominal pain (Gastrointestinal disorders) | 6 (9)
Pyrexia (General disorders) | 13 (17)
Acute sinusitis (Infections and infestations) | 9 (15)
Acute tonsillitis (Infections and infestations) | 7 (8)
Bronchitis (Infections and infestations) | 10 (17)
Nasopharyngitis (Infections and infestations) | 41 (73)
Pharyngitis (Infections and infestations) | 11 (12)
Upper respiratory tract infection (Infections and infestations) | 5 (6)
Blood cortisol decreased (Investigations) | 27 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 (69)
Heat rash (Skin and subcutaneous tissue disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the Sponsor 45 days prior to submission for publication or presentation, reveiw copies of abstracts or manuscripts for publication that report any results of the trial. The Sponsor shall have the right to reveiw and comment with respect to publications, abstracts, slides, and manuscripts and the right to reveiw and comment on the data analysis and presentation.